CLINICAL TRIAL: NCT03610581
Title: A Randomized, Double-blind, Placebo-controlled, First-in-Human, Phase 1/2a Study to Evaluate Safety, Reactogenicity and Immunogenicity of Monovalent HPV16 and HPV18 Ad26-vectored Vaccine Components and an MVA-vectored HPV16/18 Vaccine Component in Otherwise Healthy Women With HPV16 or 18 Infection of the Cervix
Brief Title: Safety, Reactogenicity and Immunogenicity of Adenovirus Serotype 26 (Ad26)- and Modified Vaccinia Ankara (MVA)-Vectored Vaccine Components in Otherwise Healthy Women With HPV16 or HPV18 Infection of the Cervix
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low enrolment and increasing COVID restrictions, following an earlier enrolment pause in April made it clear that completion of the study would not be feasible
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Collaborators: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108458; 2018-000200-41 (EudraCT Number); VAC81623HPV1002 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Results first posted 2021-11-09 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Human Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Regimen 1: Single Ad26.HPV16 or Ad26.HPV18 and MVA.HPV16/18 (Experimental): Participants will receive a dose of adenovirus serotype 26 (Ad26)-human papillomavirus (HPV)16 or HPV18 (Ad26.HPV16 or Ad26.HPV18) as prime immunization and a dose of Modified Vaccinia Ankara (MVA)-HPV16/18 (MVA.HPV16/18) as boost immunization.
  Interventions: Biological: Ad26.HPV16; Biological: Ad26.HPV18; Biological: MVA.HPV16/18
- Regimen 2: Double Ad26.HPV16 or Ad26.HPV18 and MVA.HPV16/18 (Experimental): Participants will receive a double dose of Ad26.HPV16 or Ad26.HPV18 as prime immunization and a dose of MVA.HPV16/18 as boost immunization.
  Interventions: Biological: Ad26.HPV16; Biological: Ad26.HPV18; Biological: MVA.HPV16/18
- Regimen 3: Ad26.HPV16/Ad26.HPV18 mix and MVA.HPV16/18 (Experimental): Participants will receive a mix of Ad26.HPV16/Ad26.HPV18 as prime immunization and a dose of MVA.HPV16/18 as boost immunization.
  Interventions: Biological: Ad26.HPV16; Biological: Ad26.HPV18; Biological: MVA.HPV16/18
- Control: Placebo (Placebo Comparator): Participants will receive matched placebo as prime and boost immunizations.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ad26.HPV16 — Participants will receive Ad26.HPV16 as a solution for intramuscular injection.
  Other Names: JNJ-63682918
  Arms: Regimen 1: Single Ad26.HPV16 or Ad26.HPV18 and MVA.HPV16/18; Regimen 2: Double Ad26.HPV16 or Ad26.HPV18 and MVA.HPV16/18; Regimen 3: Ad26.HPV16/Ad26.HPV18 mix and MVA.HPV16/18
Biological: Ad26.HPV18 — Participants will receive Ad26.HPV18 as a solution for intramuscular injection.
  Other Names: JNJ-63682931
  Arms: Regimen 1: Single Ad26.HPV16 or Ad26.HPV18 and MVA.HPV16/18; Regimen 2: Double Ad26.HPV16 or Ad26.HPV18 and MVA.HPV16/18; Regimen 3: Ad26.HPV16/Ad26.HPV18 mix and MVA.HPV16/18
Biological: MVA.HPV16/18 — Participants will receive MVA.HPV16/18 as a solution for intramuscular injection.
  Other Names: JNJ-65195208
  Arms: Regimen 1: Single Ad26.HPV16 or Ad26.HPV18 and MVA.HPV16/18; Regimen 2: Double Ad26.HPV16 or Ad26.HPV18 and MVA.HPV16/18; Regimen 3: Ad26.HPV16/Ad26.HPV18 mix and MVA.HPV16/18
Biological: Placebo — Participants will receive matched placebo as a solution for intramuscular injection.
  Arms: Control: Placebo

SUMMARY:
The main purpose of this study is to assess safety and reactogenicity of the 3 vaccine regimens.

DETAILED DESCRIPTION:
This study is part of a vaccine program which aims to generate a therapeutic vaccine for women with HPV types 16 or 18 infection, with a focus on early disease interception. The study consists of 3 periods: Screening period of up to 42 days (6 weeks), followed by prime and boost immunizations and follow-up visits up to 12 months after the first vaccination. Evaluation of the safety/reactogenicity of the vaccine regimens will include physical assessment by study-site personnel, participant reports on signs and symptoms and laboratory assessments following vaccinations. Immunogenicity and Virology/Histology assessments will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Must have an human papillomavirus (HPV) type 16 or 18 infection of the cervix as determined by a qualitative PCR test within 8 weeks prior to screening or at the time of screening. Available history of high-risk (HR)-HPV positivity and HPV16 or HPV18 positivity positivity will be recorded
* Must have a recent colposcopy result (with a maximum of 12 months old at screening); in case a colposcopy has not been performed before, it will be done as screening procedure
* Contraceptive (birth control) use by participants should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies
* Agrees not to donate blood until 3 months after receiving the last dose of study vaccine

Exclusion Criteria:

* In case cytology results are available, participant has current or history of high-grade squamous intraepithelial lesion (HSIL), adenocarcinoma in situ (AIS) or any high-grade vulvar, vaginal or anal intraepithelial neoplasia
* Current or history of cervical intraepithelial neoplasia (CIN)2+ or cervical cancer
* Confirmed co-infection with both HPV16 and HPV18
* History of an underlying clinically significant acute or chronic medical condition, other than infection with HPV, or physical examination findings for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Tests positive for human immunodeficiency virus (HIV) at screening
* Chronic active hepatitis B or hepatitis C infection, verified at screening by hepatitis B surface antigen or anti-hepatitis C virus antibody, respectively
* Vaginal atrophy with or without topical hormonal therapies or systemic selective estrogen receptor modulators
* Exposed to at least 1 dose of an HPV prophylactic vaccine or participant has participated in the past in another preventive or therapeutic HPV vaccine study
* Clinically significant gynecological abnormalities that could, in the judgment of the investigator, interfere with study evaluation (for example [e.g.], prolapse, myoma, fibroid, hysterectomy)
* Symptomatic vaginal or genital infection (including genital herpes) as confirmed by physician or investigator

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (12):
- United States (11):
  - Doral Medical Research, Doral, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Florida Research Center Inc., Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - University of Iowa Hospital, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Medpharmics, LLC, Metairie, Louisiana
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Columbia University Medical Center, New York, New York
  - VGR & NOCCR - Knoxville, Knoxville, Tennessee
- UZ Leuven, Leuven, Belgium

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to premature study termination, participants were only randomized and treated for Regimen 1 and Placebo. Hence, all results are reported below for Regimen 1 and Placebo only and not for Regimen 2 and 3.
Groups:
- Regimen 1: Participants received adenovirus serotype 26. human papillomavirus (Ad26.HPV)16 (Regimen 1a) or Ad26.HPV18 (Regimen 1b) at a single low dose of 5*10^10 viral particles (vp) on Day 1 followed by modified vaccinia Ankara (MVA).HPV16/18 at 2*10^8 infectious units (Inf.U) on Day 57.
- Placebo: Participants received matching placebo on Day 1 and Day 57.
Period: Overall Study
Arm/Group | Regimen 1 | Placebo
Started | 5 | 4
Vaccinated | 4 | 4
Completed | 2 | 3
Not Completed | 3 | 1
Not completed — Study terminated by sponsor | 2 | 0
Not completed — Other | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants with at least one vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen 1 | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (11.85) | 45.5 (5.69) | 43.6 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Adverse Events (AEs)
Description: Number of participants with solicited local AEs were reported. Solicited local AE's included pain/tenderness, erythema, and induration/swelling.
Time Frame: Up to 7 days after each vaccination (Up to Day 64)
Population: Full analysis set (FAS) included all participants with at least one vaccination. Here, "n (number analyzed)" is defined as participants analyzed for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 | Placebo
Number analyzed (Participants) | 5 | 4
Participants
  Post- Dose 1 | 2 | 0
  Post- Dose 2: number analyzed (Participants) | 4 | 4
  Post- Dose 2 | 1 | 0

2. Primary Outcome: Number of Participants With Solicited Systemic AEs
Description: Number of participants with solicited systemic AEs were reported. Solicited systemic AEs included headache, fatigue, myalgia, arthralgia, chills, and fever.
Time Frame: Up to 7 days after each vaccination (Up to Day 64)
Population: FAS included all participants with at least one vaccination. Here, "n (number analyzed)" is defined as participants analyzed for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 | Placebo
Number analyzed (Participants) | 5 | 4
Participants
  Post-Dose 1 | 4 | 0
  Post-Dose 2: number analyzed (Participants) | 4 | 4
  Post-Dose 2 | 1 | 0

3. Primary Outcome: Number of Participants With Unsolicited AEs
Description: Number of participants with unsolicited AEs were reported. Unsolicited AEs included all AEs for which the participant was not specifically questioned in the participant diary.
Time Frame: 28 days after each vaccination (Up to Day 85)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 | Placebo
Number analyzed (Participants) | 5 | 4
Participants
  Post-Dose 1 | 2 | 1
  Post-Dose 2: number analyzed (Participants) | 4 | 4
  Post-Dose 2 | 0 | 0

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants with SAEs were reported. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to 12 months after the first vaccination (target visit Day 366)
Population: FAS included all participants with at least one vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen 1 | Placebo
Number analyzed (Participants) | 5 | 4
Participants | 0 | 0

5. Secondary Outcome: Percentage of Participants With Human Papillomavirus (HPV)-Specific CD4+ T-cell Responses: Interferon (IFN)g+
Description: Percentage of participants with HPV-Specific CD4+ T-cell responses for IFNg+ to peptide pools were reported. Cellular immunogenicity was measured by intracellular cytokine staining (ICS), allowing characterization of individual CD4 and CD8 T cell immune responses to vaccination. The different peptide pools for HPV16 or HPV 18 were: E2, E6/E7 and combined (E2 and E6/E7 both).
Time Frame: Day 57, Day 78, Day 239, and Day 366
Population: FAS included all participants with at least one vaccination. Here, N (number of participants analyzed) is defined as participants evaluable for this outcome measure. Here, "n (number analyzed)" is defined as participants analyzed for specified category.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Regimen 1 | Placebo
Number analyzed (Participants) | 4 | 4
Percentage of participants
  Day 57: E2 | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: E2: number analyzed (Participants) | 3 | 3
  Day 78: E2 | 33.3 [0.8 to 90.6] | 0 [0 to 70.8]
  Day 239: E2: number analyzed (Participants) | 3 | 3
  Day 239: E2 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 366: E2: number analyzed (Participants) | 2 | 3
  Day 366: E2 | 0 [0 to 84.2] | 0 [0 to 70.8]
  Day 57: E6/E7 | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: E6/E7: number analyzed (Participants) | 3 | 3
  Day 78: E6/E7 | 33.3 [0.8 to 90.6] | 0 [0 to 70.8]
  Day 239: E6/E7: number analyzed (Participants) | 3 | 3
  Day 239: E6/E7 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 366: E6/E7: number analyzed (Participants) | 2 | 3
  Day 366: E6/E7 | 0 [0 to 84.2] | 0 [0 to 70.8]
  Day 57: Combined Peptide Pools | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: Combined Peptide Pools: number analyzed (Participants) | 3 | 3
  Day 78: Combined Peptide Pools | 33.3 [0.8 to 90.6] | 0 [0 to 70.8]
  Day 239: Combined Peptide Pools: number analyzed (Participants) | 3 | 3
  Day 239: Combined Peptide Pools | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 366: Combined Peptide Pools: number analyzed (Participants) | 2 | 3
  Day 366: Combined Peptide Pools | 0 [0 to 84.2] | 0 [0 to 70.8]

6. Secondary Outcome: Percentage of Participants With HPV-Specific CD4+ T-cell Responses: Interleukin (IL)2+
Description: Percentage of participants with HPV-Specific CD4+ T-cell responses for IL2+ were reported. Cellular immunogenicity was measured by intracellular cytokine staining (ICS), allowing characterization of individual CD4 and CD8 T cell immune responses to vaccination. The different peptide pools for HPV16 or HPV 18 were: E2, E6/E7 and combined (E2 and E6/E7 both).
Time Frame: Day 57, Day 78, Day 239, and Day 366
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Regimen 1 | Placebo
Number analyzed (Participants) | 4 | 4
Percentage of participants
  Day 57: E2 | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: E2: number analyzed (Participants) | 3 | 3
  Day 78: E2 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 239: E2: number analyzed (Participants) | 3 | 3
  Day 239: E2 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 366: E2: number analyzed (Participants) | 2 | 3
  Day 366: E2 | 0 [0 to 84.2] | 0 [0 to 70.8]
  Day 57: E6/E7 | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: E6/E7: number analyzed (Participants) | 3 | 3
  Day 78: E6/E7 | 33.3 [0.8 to 90.6] | 0 [0 to 70.8]
  Day 239: E6/E7: number analyzed (Participants) | 3 | 3
  Day 239: E6/E7 | 33.3 [0.8 to 90.6] | 0 [0 to 70.8]
  Day 336: E6/E7: number analyzed (Participants) | 2 | 3
  Day 336: E6/E7 | 0 [0 to 84.2] | 0 [0 to 70.8]
  Day 57: Combined Peptide Pools | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: Combined Peptide Pools: number analyzed (Participants) | 3 | 3
  Day 78: Combined Peptide Pools | 33.3 [0.8 to 90.6] | 0 [0 to 70.8]
  Day 239: Combined Peptide Pools: number analyzed (Participants) | 3 | 3
  Day 239: Combined Peptide Pools | 33.3 [0.8 to 90.6] | 0 [0 to 70.8]
  Day 366: Combined Peptide Pools: number analyzed (Participants) | 2 | 3
  Day 366: Combined Peptide Pools | 0 [0 to 84.2] | 0 [0 to 70.8]

7. Secondary Outcome: Percentage of Participants With HPV-Specific CD4+ T-cell Responses: Tumor Necrosis Factor (TNF)a+
Description: Percentage of participants with HPV-Specific CD4+ T-cell responses for TNF a+ were reported. Cellular immunogenicity was measured by intracellular cytokine staining (ICS), allowing characterization of individual CD4 and CD8 T cell immune responses to vaccination. The different peptide pools for HPV16 or HPV 18 were: E2, E6/E7 and combined (E2 and E6/E7 both).
Time Frame: Day 57, Day 78, Day 239, and Day 366
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Regimen 1 | Placebo
Number analyzed (Participants) | 4 | 4
Percentage of participants
  Day 57: E2 | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: E2: number analyzed (Participants) | 3 | 3
  Day 78: E2 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 239: E2: number analyzed (Participants) | 3 | 3
  Day 239: E2 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 366: E2: number analyzed (Participants) | 2 | 3
  Day 366: E2 | 0 [0 to 84.2] | 0 [0 to 70.8]
  Day 57: E6/E7 | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: E6/E7: number analyzed (Participants) | 3 | 3
  Day 78: E6/E7 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 239: E6/E7: number analyzed (Participants) | 3 | 3
  Day 239: E6/E7 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 366: E6/E7: number analyzed (Participants) | 2 | 3
  Day 366: E6/E7 | 0 [0 to 84.2] | 0 [0 to 70.8]
  Day 57: Combined Peptide Pools | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: Combined Peptide Pools: number analyzed (Participants) | 3 | 3
  Day 78: Combined Peptide Pools | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 239: Combined Peptide Pools: number analyzed (Participants) | 3 | 3
  Day 239: Combined Peptide Pools | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 366: Combined Peptide Pools: number analyzed (Participants) | 2 | 3
  Day 366: Combined Peptide Pools | 0 [0 to 84.2] | 0 [0 to 70.8]

8. Secondary Outcome: Percentage of Participants With HPV-Specific CD8+ T-cell Responses: IFNg+
Description: Percentage of participants with HPV-Specific CD8+ T-cell responses for IFNg+ were reported. Cellular immunogenicity was measured by intracellular cytokine staining (ICS), allowing characterization of individual CD4 and CD8 T cell immune responses to vaccination. The different peptide pools for HPV16 or HPV 18 were: E2, E6/E7 and combined (E2 and E6/E7 both).
Time Frame: Day 57, Day 78, Day 239, and Day 366
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Regimen 1 | Placebo
Number analyzed (Participants) | 4 | 4
Percentage of participants
  Day 57: E2 | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: E2: number analyzed (Participants) | 3 | 3
  Day 78: E2 | 100 [29.2 to 100] | 0 [0 to 70.8]
  Day 239: E2: number analyzed (Participants) | 3 | 3
  Day 239: E2 | 66.7 [9.4 to 99.2] | 0 [0 to 70.8]
  Day 366: E2: number analyzed (Participants) | 2 | 3
  Day 366: E2 | 50 [1.3 to 98.7] | 0 [0 to 70.8]
  Day 57: E6/E7 | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: E6/E7: number analyzed (Participants) | 3 | 3
  Day 78: E6/E7 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 239: E6/E7: number analyzed (Participants) | 3 | 3
  Day 239: E6/E7 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 366: E6/E7: number analyzed (Participants) | 2 | 3
  Day 366: E6/E7 | 0 [0 to 84.2] | 0 [0 to 70.8]
  Day 57: Combined Peptide Pools | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: Combined Peptide Pools: number analyzed (Participants) | 3 | 3
  Day 78: Combined Peptide Pools | 100 [29.2 to 100] | 0 [0 to 70.8]
  Day 239: Combined Peptide Pools: number analyzed (Participants) | 3 | 3
  Day 239: Combined Peptide Pools | 66.7 [9.4 to 99.2] | 0 [0 to 70.8]
  Day 366: Combined Peptide Pools: number analyzed (Participants) | 2 | 3
  Day 366: Combined Peptide Pools | 50 [1.3 to 98.7] | 0 [0 to 70.8]

9. Secondary Outcome: Percentage of Participants With HPV-Specific CD8+ T-cell Responses: IL2+
Description: Percentage of participants with HPV-Specific CD8+ T-cell responses for IL2+ were reported. Cellular immunogenicity was measured by intracellular cytokine staining (ICS), allowing characterization of individual CD4 and CD8 T cell immune responses to vaccination. The different peptide pools for HPV16 or HPV 18 were: E2, E6/E7 and combined (E2 and E6/E7 both).
Time Frame: Day 57, Day 78, Day 239, and Day 366
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Regimen 1 | Placebo
Number analyzed (Participants) | 4 | 4
Percentage of participants
  Day 57: E2 | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: E2: number analyzed (Participants) | 3 | 3
  Day 78: E2 | 66.7 [9.4 to 99.2] | 0 [0 to 70.8]
  Day 239: E2: number analyzed (Participants) | 3 | 3
  Day 239: E2 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 366: E2: number analyzed (Participants) | 2 | 3
  Day 366: E2 | 50 [1.3 to 98.7] | 0 [0 to 70.8]
  Day 57: E6/E7 | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: E6/E7: number analyzed (Participants) | 3 | 3
  Day 78: E6/E7 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 239: E6/E7: number analyzed (Participants) | 3 | 3
  Day 239: E6/E7 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 366: E6/E7: number analyzed (Participants) | 2 | 3
  Day 366: E6/E7 | 0 [0 to 84.2] | 0 [0 to 70.8]
  Day 57: Combined Peptide Pools | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: Combined Peptide Pools: number analyzed (Participants) | 3 | 3
  Day 78: Combined Peptide Pools | 66.7 [9.4 to 99.2] | 0 [0 to 70.8]
  Day 239: Combined Peptide Pools: number analyzed (Participants) | 3 | 3
  Day 239: Combined Peptide Pools | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 366: Combined Peptide Pools: number analyzed (Participants) | 2 | 3
  Day 366: Combined Peptide Pools | 50 [1.3 to 98.7] | 0 [0 to 70.8]

10. Secondary Outcome: Percentage of Participants With HPV-Specific CD8+ T-cell Responses: TNFa+
Description: Percentage of participants with HPV-Specific CD8+ T-cell responses for TNFa+ were reported. Cellular immunogenicity was measured by intracellular cytokine staining (ICS), allowing characterization of individual CD4 and CD8 T cell immune responses to vaccination. The different peptide pools for HPV16 or HPV 18 were: E2, E6/E7 and combined (E2 and E6/E7 both).
Time Frame: Day 57, Day 78, Day 239, and Day 366
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Regimen 1 | Placebo
Number analyzed (Participants) | 4 | 4
Percentage of participants
  Day 57: E2 | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: E2: number analyzed (Participants) | 3 | 3
  Day 78: E2 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 239: E2: number analyzed (Participants) | 3 | 3
  Day 239: E2 | 33.3 [0.8 to 90.6] | 0 [0 to 70.8]
  Day 366: E2: number analyzed (Participants) | 2 | 3
  Day 366: E2 | 0 [0 to 84.2] | 0 [0 to 70.8]
  Day 57: E6/E7 | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: E6/E7: number analyzed (Participants) | 3 | 3
  Day 78: E6/E7 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 239: E6/E7: number analyzed (Participants) | 3 | 3
  Day 239: E6/E7 | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 366: E6/E7: number analyzed (Participants) | 2 | 3
  Day 366: E6/E7 | 0 [0 to 84.2] | 0 [0 to 70.8]
  Day 57: Combined Peptide Pools | 0 [0 to 60.2] | 0 [0 to 60.2]
  Day 78: Combined Peptide Pools: number analyzed (Participants) | 3 | 3
  Day 78: Combined Peptide Pools | 0 [0 to 70.8] | 0 [0 to 70.8]
  Day 239: Combined Peptide Pools: number analyzed (Participants) | 3 | 3
  Day 239: Combined Peptide Pools | 33.3 [0.8 to 90.6] | 0 [0 to 70.8]
  Day 366: Combined Peptide Pools: number analyzed (Participants) | 2 | 3
  Day 366: Combined Peptide Pools | 0 [0 to 84.2] | 0 [0 to 70.8]

ADVERSE EVENTS:
Time Frame: Up to 12 months after the first vaccination (target visit Day 366)
Description: Full analysis set (FAS) included all participants with at least one vaccination.
Arm/Group | Regimen 1 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 2/5 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 (N=5) | Placebo (N=4)
Increased Tendency to Bruise (Blood and lymphatic system disorders) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
As the study was terminated prematurely, the Sponsor performed a limited analysis on the available data to meet the requirement for reporting the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT03610581/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT03610581/SAP_001.pdf